CLINICAL TRIAL: NCT02910102
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled Crossover Study Evaluating the Effect of RVT-101 on Gait and Balance in Subjects With Alzheimer's Disease, Dementia With Lewy Bodies, or Parkinson's Disease Dementia
Brief Title: Study Evaluating Intepirdine (RVT-101) on Gait and Balance in Subjects With Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Axovant Sciences Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sio Gene Therapies (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVT-101-2003
Record Dates: First submitted 2016-09-16; First posted 2016-09-21 (Estimated); Results first posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2019-01

CONDITIONS: Alzheimer's Disease; Dementia With Lewy Bodies; Parkinson's Disease Dementia
Keywords: RVT-101; intepirdine; Alzheimer's disease; Dementia with Lewy bodies; Lewy body dementia; Parkinson's Disease Dementia
MeSH Terms: conditions — Alzheimer Disease; Lewy Body Disease | interventions — 3-benzenesulfonyl-8-piperazin-1-ylquinoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence AB (Other): RVT-101 35 mg in Period II and Placebo in Period IV
  Interventions: Drug: RVT-101 35 mg; Drug: Placebo
- Sequence BA (Other): Placebo in Period II and RVT-101 35 mg in Period IV
  Interventions: Drug: RVT-101 35 mg; Drug: Placebo

INTERVENTIONS:
Drug: RVT-101 35 mg — RVT-101 once daily, oral, 35-mg tablets
Drug: Placebo — Placebo once daily, oral

SUMMARY:
This study seeks to evaluate the effect of intepirdine (RVT-101) on gait and balance in patients with Alzheimer's Disease, Dementia with Lewy Bodies or Parkinson's Disease Dementia.

DETAILED DESCRIPTION:
To assess the effect of intepirdine (RVT-101) versus placebo on quantitative and qualitative gait and balance parameters.

Each subject will be randomized 1:1 to one of the following sequences:

Sequence 1: AB = RVT-101 35 mg during the early treatment period and Placebo during the late treatment period

Sequence 2: BA = Placebo during the early treatment period and RVT-101 35 mg during the late treatment period

Treatment A = RVT-101 35 mg once daily.

Treatment B = Placebo once daily.

ELIGIBILITY:
Key Inclusion Criteria:

Male or female subject with a clinical diagnosis of Alzheimer's disease (AD), dementia with Lewy bodies (DLB), or Parkinson's disease dementia (PDD).

Mini Mental State Examination score 14 to 26 Gait impairment, as assessed by history gathered by the clinical investigator and quantitative measurements Subjects must be on stable background acetylcholinesterase inhibitor therapy

Key Exclusion Criteria:

History and/or evidence of any other CNS disorder that could be interpreted as a cause of dementia (in the opinion of the investigator) Any clinically relevant concomitant disease which, in the opinion of the investigator, makes the subject unsuitable for inclusion in the study.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilise Lombardo, MD, Study Chair — Axovant Sciences, Inc., Senior VP Clinical Research
Locations (11):
- United States (11):
  - US101, Phoenix, Arizona
  - US118, Simi Valley, California
  - US117, Temecula, California
  - US115, Boca Raton, Florida
  - US109, Hallandale, Florida
  - US116, Miami, Florida
  - US108, Pensacola, Florida
  - US106, Columbus, Georgia
  - US107, Indianapolis, Indiana
  - US102, Ann Arbor, Michigan
  - US111, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 68 participants signed consent and were screened for participation. Of these, 40 entered a 2-week single-blind placebo run-in period with treatment with placebo qd. Subjects were allowed to re-screen if they failed the initial screening assessments. All subjects deemed eligible following run-in were randomized to a treatment group.
Groups:
- Sequence 1: AB: RVT-101 35 mg: once daily, oral, 35-mg tablets in Period II
  Placebo in Period IV
- Sequence 2: BA: Placebo: once daily, oral, matching tablets in Period II
  RVT-101 35 mg: once daily, oral, 35-mg tablets in Period IV
Period: Overall Study
Arm/Group | Sequence 1: AB | Sequence 2: BA
Started | 21 | 17
Safety Population (The Safety population included subjects who took at least 1 dose of double-blind study drug) | 21 | 17
Intent to Treat (ITT) Population (Subjects took at least 1 dose of DB study drug and had at least 1 post-baseline assessment) | 21 | 17
Per-Protocol Population (Subjects in the ITT population who had no major protocol violations) | 20 | 17
Completed (Subjects in the ITT population who completed the study) | 21 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1: AB | Sequence 2: BA | Total
Number analyzed (Participants) | 21 | 17 | 38
Age, Continuous [Mean (Full Range); unit: years] | 76.0 [68 to 86] | 73.8 [60 to 83] | 75.0 [60 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 4 | 18
  Male | 7 | 13 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 14 | 11 | 25
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 20 | 15 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Full Range); unit: kg/m^2] | 27.312 [19.23 to 45.59] | 25.898 [16.01 to 34.57] | 26.680 [16.01 to 45.59]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Gait Speed (cm/Sec) Measurements From Baseline to the End of Each Double-blind Treatment Period Based on Computerized Gait Assessment Tools.
Description: Change from baseline in gait speed (cm/sec) measured on an electronic walkway system under single task trial condition (meaning walking only) at the end of each two-week treatment period
Time Frame: Baseline, 2 weeks
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: cm/sec
Groups:
- RVT-101 35 mg: Subjects who dosed with RVT-101 in both sequences (AB and BA) are included in this analysis
- Placebo: Subjects who dosed with Placebo in both sequences (AB and BA) are included in this analysis
Arm/Group | RVT-101 35 mg | Placebo
Number analyzed (Participants) | 36 | 37
cm/sec | -0.43 (1.845) | 1.47 (1.874)
Statistical Analysis 1: Comparison: RVT-101 35 mg vs Placebo; Test type: Superiority; p = 0.3565, Mixed Models Analysis — The threshold for statistical significance was p=0.05; Each co-primary endpoint was tested at two-sided 5% level of significance, with no adjustments for multiplicity; Mean Difference (Final Values) = -1.90, 95% CI 2-sided [-6.04 to 2.23]

2. Primary Outcome: Change in Gait Measurements (cm/Sec) Under Dual Task Condition From Baseline to the End of Each Double-blind Treatment Period Based on Computerized Gait Assessment Tools.
Description: Change from baseline in gait speed (cm/sec) measured on an electronic walkway system under dual task trial condition (meaning walking while performing another task) at the end of each two-week treatment period.
Time Frame: Baseline, 2 weeks
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: cm/sec
Groups:
- RVT-101 35 mg: RVT-101 35 mg: once daily, oral
  Subjects who dosed with RVT-101 in both sequences (AB and BA) are included in this analysis
Arm/Group | RVT-101 35 mg | Placebo
Number analyzed (Participants) | 36 | 37
cm/sec | 1.46 (1.517) | 1.63 (1.518)
Statistical Analysis 1: Comparison: RVT-101 35 mg vs Placebo; Test type: Superiority; p = 0.9220, Mixed Models Analysis — The threshold for statistical significance was p=0.05; Each co-primary endpoint was tested at two-sided 5% level of significance, with no adjustments for multiplicity; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-3.73 to 3.38]

ADVERSE EVENTS:
Time Frame: Screening through post-treatment (Up to 16 Weeks)
Groups:
- RVT-101 35 mg: Subjects who dosed with RVT-101 in both sequences (AB and BA) are included
- Placebo: Subjects who dosed with Placebo in both sequences (AB and BA) are included
- Screening Period: Participants screened (0-4 weeks) prior to entering to the first dose of single-blind study medication (ie, prior to the Run-In period)
- Run-In Period: Placebo: once daily, oral, pill manufactured to match RVT-101 35 mg tablet (for 2 weeks)
- RVT-101 Post-Treatment; Placebo Post-Treatment: Subjects reported adverse events after completing the treatment period. The Post-Treatment period - defined as up to 17 days post-last-dose
Arm/Group | RVT-101 35 mg | Placebo | Screening Period | Run-In Period | RVT-101 Post-Treatment | Placebo Post-Treatment
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38 | 0/68 | 0/40 | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38 | 0/68 | 0/40 | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38 | 0/68 | 0/40 | 0/38 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All proposed manuscripts, publications or abstracts must be reviewed and approved by the Sponsor 60 days prior to submission for publication. All confidential information identified by the Sponsor must be deleted prior to submission.

DOCUMENTS (2):
  • Study Protocol (2017-02-07): https://cdn.clinicaltrials.gov/large-docs/02/NCT02910102/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT02910102/SAP_001.pdf